CLINICAL TRIAL: NCT03050346
Title: Breathing-Induced Myocardial Oxygenation Reserve - Pilot Study (B-MORE-Pilot)
Brief Title: Breathing-Induced Myocardial Oxygenation Reserve
Acronym: B-MORE-Pilot
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University Hospital Heidelberg (Other); Groote Schuur Hospital (Unknown); King's College London (Other); University of Wisconsin, Madison (Other); Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Chief, Cardiovascular Imaging, McGill University Health Centre, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 15-398-MUHC
Record Dates: First submitted 2017-02-08; First posted 2017-02-10 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Coronary Artery Disease
Keywords: Magnetic Resonance Imaging; Coronary Artery Disease; Apnea; Hyperventilation; BOLD; Breathing Maneuvers; Myocardial Oxygenation
MeSH Terms: conditions — Coronary Artery Disease; Apnea; Hyperventilation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CAD patients: Consecutive patients scheduled for a coronary angiography on the basis of cardiac symptoms and a test positive for inducible coronary ischemia, who are affected by one-vessel or two-vessel CAD at the time of the OS-CMR with breathing maneuvers (HVBH).
- Healthy subjects: Subjects without current or pre-existing cardiovascular and lung disease and absence of medication with cardiovascular effects.

SUMMARY:
This is a clinical trial to test the clinical feasibility and safety of a novel CMR protocol, combined with a specific breathing maneuver to identify myocardial regions exposed to severe coronary artery stenosis.

DETAILED DESCRIPTION:
This is a clinical trial to test the clinical feasibility and safety of a novel CMR protocol. It aims to investigate a new Cardiovascular Magnetic Resonance (CMR) technique, called oxygenation-sensitive CMR (OS-CMR).

OS-CMR is a T2*-sensitive CMR sequence based on the so-called blood-oxygen-level-dependent (BOLD) effect. Because de-oxygenated hemoglobin acts as an endogenous paramagnetic contrast agent, the signal intensity (SI) in OS-CMR images is linearly correlated with hemoglobin oxygenation in the tissue. An increase in deoxyhemoglobin results in an drop in SI in OS-CMR images, while an increase in tissue oxygenation results in an increase in SI.

Therefore, OS-CMR has been found capable of assessing myocardial oxygenation and is being increasingly used to identify the vascular response of the coronary circulation to different stimuli.

Very recently, OS-CMR was used to identify the coronary vascular response to specific breathing maneuvers. Specifically, a marked increase of myocardial oxygenation was observed during a long breath-hold following a 60s period of hyperventilation. The combination of these two maneuvers appear to induce consistent and detectable changes of myocardial oxygenation, based on CO2-mediated coronary vasoconstriction and vasodilation, while being well tolerated by participants.

In this study, the investigators will use breathing maneuvers as coronary vasoactive stimuli to assess the myocardial oxygenation changes induced by such maneuvers with OS-CMR.

The investigators aim to assess if the breathing-induced relative increase of myocardial oxygenation (Breathing-induced Myocardial Oxygenation REserve, B-MORE) in a coronary territory is clinically feasible to serve as a marker for the severity of coronary artery stenosis.

Moreover, the investigators will assess the feasibility and safety of OS-CMR with breathing maneuvers in patients with suspected coronary artery disease in a multi-center setting.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Informed consent as documented by signature (Appendix Informed Consent Form)
* Indication for invasive coronary angiography based on symptoms and a test positive for inducible coronary ischemia
* One-vessel or two-vessel CAD at coronary angiography (For healthy volunteers: absence of current or pre-existing cardiovascular and lung disease and absence of medication with cardiovascular effects)

Exclusion Criteria:

* General MRI contraindications (i.e pacemakers, defibrillating wires, implanted defibrillators, intracranial aneurysm clips, metallic foreign bodies in the eyes, knowledge or suspicion of pregnancy)
* Acute Coronary Syndrome (ACS) or other acute cardiac injury within 4 weeks
* Previous myocardial infarction, percutaneous coronary intervention or coronary artery bypass surgery
* Hemodynamically unstable conditions
* Significant or uncontrolled arrhythmias
* Lack of ability to follow commands
* Vasoactive medication (e.g. nitro or ß blockers) or nutrition with caffeine (coffee, tea, cocoa, chocolate, "energy drink") during the 12 h before the exam
* Non-ischemic cardiomyopathy
* Severe Pulmonary Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients scheduled for a coronary angiography on the basis of cardiac symptoms and a test positive for inducible coronary ischemia, who show one-vessel or two-vessel CAD at coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-01; Primary Completion 2019-06 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
Comparison of myocardial oxygenation signal intensity changes (OS-SI) changes between healthy and post-stenotic myocardium during OS-CMR with breathing-maneuvers in CAD patients. | OS-CMR with breathing maneuvers will last about 5-10 minutes
  Myocardial oxygenation signal intensity changes (OS-SI) changes between healthy and post-stenotic myocardium during OS-CMR with breathing-maneuvers

SECONDARY OUTCOMES:
Relationship between OS-SI changes during OS-CMR with breathing-maneuvers and Fractional Flow Reserve (FFR) measurements in CAD patients | OS-CMR with breathing maneuvers will last about 5-10 minutes
  Myocardial oxygenation signal intensity changes (OS-SI) changes during OS-CMR with breathing-maneuvers and its relation to Fractional Flow Reserve (FFR) measurements
Relationship between OS-SI changes during OS-CMR with breathing-maneuvers and Quantitative Coronary Angiography (QCA) measurements in CAD patients | OS-CMR with breathing maneuvers will last about 5-10 minutes
  Myocardial oxygenation signal intensity changes (OS-SI) changes during OS-CMR with breathing-maneuvers and its relation to Quantitative Coronary Angiography (QCA) measurements
Presence of side effects during OS-CMR with breathing maneuvers | OS-CMR with breathing maneuvers will last about 5-10 minutes
  side effects experienced by the participants during breathing maneuvers
Clinical feasibility of OS-CMR with breathing maneuvers | OS-CMR with breathing maneuvers will last about 5-10 minutes
  Number of participants who voluntarily stopped the maneuver prior to completion and scan time of the image acquisition protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Friedrich, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (6):
- University of Wisconsin, Madison, Wisconsin, United States
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
- University Hospital Heidelberg, Heidelberg, Germany
- Groote Schuur Hospital, Cape Town, South Africa
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Friedrich MG, Niendorf T, Schulz-Menger J, Gross CM, Dietz R. Blood oxygen level-dependent magnetic resonance imaging in patients with stress-induced angina. Circulation. 2003 Nov 4;108(18):2219-23. doi: 10.1161/01.CIR.0000095271.08248.EA. Epub 2003 Oct 13. PMID 14557359
- [Background] Arnold JR, Karamitsos TD, Bhamra-Ariza P, Francis JM, Searle N, Robson MD, Howells RK, Choudhury RP, Rimoldi OE, Camici PG, Banning AP, Neubauer S, Jerosch-Herold M, Selvanayagam JB. Myocardial oxygenation in coronary artery disease: insights from blood oxygen level-dependent magnetic resonance imaging at 3 tesla. J Am Coll Cardiol. 2012 May 29;59(22):1954-64. doi: 10.1016/j.jacc.2012.01.055. PMID 22624835
- [Background] Friedrich MG, Karamitsos TD. Oxygenation-sensitive cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2013 May 24;15(1):43. doi: 10.1186/1532-429X-15-43. PMID 23706167
- [Background] Luu JM, Friedrich MG, Harker J, Dwyer N, Guensch D, Mikami Y, Faris P, Hare JL. Relationship of vasodilator-induced changes in myocardial oxygenation with the severity of coronary artery stenosis: a study using oxygenation-sensitive cardiovascular magnetic resonance. Eur Heart J Cardiovasc Imaging. 2014 Dec;15(12):1358-67. doi: 10.1093/ehjci/jeu138. Epub 2014 Aug 7. PMID 25104812
- [Background] Guensch DP, Fischer K, Flewitt JA, Friedrich MG. Impact of intermittent apnea on myocardial tissue oxygenation--a study using oxygenation-sensitive cardiovascular magnetic resonance. PLoS One. 2013;8(1):e53282. doi: 10.1371/journal.pone.0053282. Epub 2013 Jan 3. PMID 23301055
- [Background] Guensch DP, Fischer K, Flewitt JA, Yu J, Lukic R, Friedrich JA, Friedrich MG. Breathing manoeuvre-dependent changes in myocardial oxygenation in healthy humans. Eur Heart J Cardiovasc Imaging. 2014 Apr;15(4):409-14. doi: 10.1093/ehjci/jet171. Epub 2013 Sep 27. PMID 24078154
- [Background] Fischer K, Guensch DP, Friedrich MG. Response of myocardial oxygenation to breathing manoeuvres and adenosine infusion. Eur Heart J Cardiovasc Imaging. 2015 Apr;16(4):395-401. doi: 10.1093/ehjci/jeu202. Epub 2014 Oct 21. PMID 25336541
- [Background] Neill WA, Hattenhauer M. Impairment of myocardial O2 supply due to hyperventilation. Circulation. 1975 Nov;52(5):854-8. doi: 10.1161/01.cir.52.5.854. PMID 1175266
- [Background] Sueda S, Saeki H, Otani T, Ochi N, Kukita H, Kawada H, Matsuda S, Uraoka T. Investigation of the most effective provocation test for patients with coronary spastic angina: usefulness of accelerated exercise following hyperventilation. Jpn Circ J. 1999 Feb;63(2):85-90. doi: 10.1253/jcj.63.85. PMID 10084369
- [Background] Nakao K, Ohgushi M, Yoshimura M, Morooka K, Okumura K, Ogawa H, Kugiyama K, Oike Y, Fujimoto K, Yasue H. Hyperventilation as a specific test for diagnosis of coronary artery spasm. Am J Cardiol. 1997 Sep 1;80(5):545-9. doi: 10.1016/s0002-9149(97)00419-0. PMID 9294979
- [Background] Chauhan A, Mullins PA, Taylor G, Petch MC, Schofield PM. Effect of hyperventilation and mental stress on coronary blood flow in syndrome X. Br Heart J. 1993 Jun;69(6):516-24. doi: 10.1136/hrt.69.6.516. PMID 8343318